CLINICAL TRIAL: NCT02380417
Title: Paravertebral Catheter Use for Postoperative Pain Control in Patients After Lung Transplant Surgery: A Prospective Observational Study
Brief Title: Paravertebral Catheter for Lung Transplant
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1309M42821
Record Dates: First submitted 2015-02-02; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-02

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Ropivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Single lung transplant paravertebral catheter placement: Those patients who underwent single lung transplant either right or left.
  Interventions: Procedure: paravertebral catheter placement; Drug: 0.2% ropivacaine; Device: Elastomeric pump
- bilateral lung transplant paravertebral catheter placement: those patients who underwent bilateral lung transplantation
  Interventions: Procedure: paravertebral catheter placement; Drug: 0.2% ropivacaine; Device: Elastomeric pump

INTERVENTIONS:
Procedure: paravertebral catheter placement — a thoracic paravertebral catheter was placed and connected to an elastomeric pump with a continuous infusion of 0.2% ropivacaine
Drug: 0.2% ropivacaine — 0.2% ropivacaine was infused through the elastomeric device
Device: Elastomeric pump — An elastomeric pump was connected to the paravertebral catheter

SUMMARY:
This is a prospective observational trial of patient undergoing lung transplantation who have a thoracic paravertebral catheter(s) placed for postoperative pain control. Patients pain scores and opioid use were evaluated for 7 days after placement as well as any complications, opioid adverse events, and length of stay.

DETAILED DESCRIPTION:
Following approval of the University of Minnesota Institutional Review Board, 33 consecutive adult patients (≥ 18 years of age) were observed from October 2013 to December 2014 who underwent either single or bilateral lung transplantation and received a continuous paravertebral block. The paravertebral catheters were placed within 1-2 day postoperatively in the intensive care unit. If the patient was too hemodynamically unstable or too critically ill to be placed in lateral decubitus position, the placement of the catheter was delayed or in some cases not performed (these patients were not included in study) They were placed via an in plane transverse technique. The ultrasound was placed on the patient's back at the T8-9 level with probe in transverse orientation. Then a 17-gauge tuohy needle was advanced lateral to medial in plane until beneath the transverse process upon which a test dose of 3-5 mL of 1.5% lidocaine with 1:200,000 epinephrine was injected to see adequate spread. The catheter was then fed 1 centimeter past the tip of the tuohy needle and needle was withdrawn. All catheters were confirmed to be in correct position with real time local anesthetic injection and secured with skin glue and occlusive dressing. Each was performed with the patient in the left lateral decubitus position for the right catheter and right lateral decubitus position for the left catheter. The paravertebral catheters remained in place for up to seven days postoperatively in unilateral lung transplants and up to ten days postoperatively in bilateral lung transplants. During that time an infusion of 0.2% ropivacaine was infused at a rate of 0.2-0.25 ml/kg/hour through an elastomeric pump (ON Q Halyard Health).

The outcome measured were minimal and maximum pain scores from the first 7 days post paravertebral catheter placement (rated on an 11-point numeric rating scale; 0=no pain, 10=worst pain imaginable). The acute pain Nurse Practitioners, bedside nurses, or acute pain anesthesiology residents collected the pain scores. Additional outcomes of interest included postsurgical opioid use through postsurgical day 7, and length of hospital stay. Patients were asked daily if they experienced nausea/vomiting, however, Nursing notes and physician progress notes were also evaluated if patients experienced any adverse events or nausea and vomiting. Demographics such as age and weight were recorded in addition to length of surgery and time spent in the hospital before discharge.

ELIGIBILITY:
Inclusion Criteria:

* lung transplant
* clamshell incision
* received paravertebral catheter within 2 days of surgery

Exclusion Criteria:

* non english speaking
* remained intubated for greater than 3 days postoperatively
* midline incision
* allergy to local anesthetics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who presented for a lung transplant and had a clamshell incision either single or bilateral.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Maximal Pain score | each post catheter day from postoperative day 1 to day 7
  VAS pain scores assessed by bedside nurse on 0-10 scale which is maximum felt

SECONDARY OUTCOMES:
Minimal Pain score | each post catheter day from post operative day 1 to day 7
  VAS pain scores assessed by bedside nurse on 0-10 scale which is minimum felt
total opioid use | each post catheter day from postoperative day 1 to day 7
  opioids were normalized to milligrams of IV morphine
length of stay | from end of surgery evaluated until patient left hospital with expected average up to 3 weeks
  participants followed for duration of stay expected average 3 weeks
number of patients with nausea in the postoperative period | from day of surgery evaluated up to post catheter day 7